CLINICAL TRIAL: NCT06730074
Title: A Novel Robotic System for Motor-cognitive Exercise for Patients With Parkinson's Disease
Acronym: PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adi Negev-Nahalat Eran (Other)
Responsible Party: Principal Investigator, Ilanit Baum-Cohen, Occupational Therapist, Adi Negev-Nahalat Eran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0005-NGV-24
Record Dates: First submitted 2024-10-24; First posted 2024-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson-disease; SAR; Rehabilitation; Motor-Cognitive; PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study will be conducted with 15 PD patients, aged 50-75
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamified rehabilitation system involving robot for individuals with Parkinson's (Experimental): We will run a robotic exercise game with 15 PD patients who will use the system in a sitting position. Each patient will use the system 5 times, each time for 30 min. Principles of effective rehabilitation practice such as repetitive practice, goal-oriented practice, variable difficulty, rhythmic cueing, and social interaction are implemented in our design
  Interventions: Device: Using a gamified rehabilitation system in a sitting position involving robots and music for the benefit of individuals with Parkinson's disease (PD)

INTERVENTIONS:
Device: Using a gamified rehabilitation system in a sitting position involving robots and music for the benefit of individuals with Parkinson's disease (PD) — This is the first socially assistive robotic platform developed specifically for people with PD. If successful, this platform could be incorporated into the clinical toolbox at Adi Negev and other centres.

SUMMARY:
The objective of this study is to test a gamified rehabilitation system in a sitting position involving robots and music for the benefit of individuals with Parkinson's disease (PD). This pilot experiment will involve the collection of both subjective user evaluation measures and objective motor and cognitive measures.

DETAILED DESCRIPTION:
Participants & Protocol:

Recruitment: Advertising ads in movement disorders units in hospitals and medical centers in the south, as well as through the help of the Parkinson's Association.

The study will be conducted with 15 PD patients, aged 50-75, at the Adi Negev Clinic. Each patient will use the robotic system five times, with each session lasting 30 minutes. The intervention plan incorporates principles of effective rehabilitation practice, including repeated practice, goal-oriented practice, variable difficulty, rhythmic cueing, and social interaction. Before the research begins, participants will sign an informed consent form.

Baseline and Pre-Post Tests:

Assessments including the MoCA, demographic data, clinical data, Color Trails Test (CTT), motor UPDRS, Box & Blocks Test, and Cognitive Reserve Index Questionnaire (CRIq) will be collected before the first session by an occupational or physical therapist. After the fifth session, post-intervention assessments will include motor UPDRS, Box & Blocks Test, CTT, System Usability Scale (SUS), Intrinsic Motivation Inventory (IMI), and a satisfaction questionnaire.

Hypothesis:

It is hypothesized that motor and cognitive training using the robots will improve the patients' clinical symptoms, as evidenced by pre-post test results.

Novelty & Impact:

This is the first socially assistive robotic platform developed specifically for people with PD. If successful, this platform could be incorporated into the clinical toolbox at Adi Negev and other centres. Additionally, this study will be the first to use the Cognitive Reserve Index Questionnaire (CRIq) in Hebrew for people with PD. The potential impact of this project is twofold: testing a new rehabilitation tool and a screening tool for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form
* Men and women in ages 50-75
* Hebrew speakers
* Have Idiopathic Parkinson's disease
* Hoehn and Yahr 3 and below
* Moca test 23 and above

Exclusion Criteria:

* Patients with Parkinson's plus syndromes
* PD patients who suffer from unrelated neurological symptoms.
* Orthopedic problems of the upper limb
* Recent surgery conducted on the upper limb
* Uncorrected vision problems
* Uncorrected severe hearing loss

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
level of engagement | 2 Mon
  We will ask participants to rate their perceived level of engagement with the platform.

SECONDARY OUTCOMES:
improvement in UPDRS | 4 Mon
  We will perform post-intervention assessments which include motor UPDRS (Unified Parkinson Disease Rating Scale)
improvement in fine motor coordination | 4 Mon
  We will perform post-intervention assessments which include Box and Blocks Test for fine motor coordination.
improvement in CTT (Color Trail Test) | 4 Mon
  We will perform post-intervention assessments which include CTT (Color Trail Test) for executive functions.
Testing the usability of use of the system | 4 Mon
  We will perform post-intervention assessments which include System Usability Scale (SUS).
Measuring the motivation to use the system | 4 Mon
  We will perform post-intervention assessments which include the Intrinsic Motivation Inventory (IMI).

CONTACTS AND LOCATIONS:
Locations (1):
- Adi Negev, Ofakim, South, Israel